CLINICAL TRIAL: NCT04061720
Title: Identifying Effective Treatment for Veterans Unwilling to Quit Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NURA-009-18F
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Tobacco Dependence; Veterans
Keywords: Tobacco dependence; Clinical Trial; Veterans
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced Chronic Care (Experimental): Enhanced Chronic Care provides ongoing, phone-based motivational interventions and interpersonal support to promote readiness to quit, with facilitated access to evidence-based smoking treatment.
  Interventions: Behavioral: Enhanced Chronic Care
- Standard Care (Active Comparator): Standard Care provides phone-based brief advice to quit once per year.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Enhanced Chronic Care — Enhanced Chronic Care involves four chronic care calls per year. Enhanced Chronic Care is designed to help participants explore their goals and concerns with regard to smoking, engage in a nondirective, supportive, motivational interventions, and provide information about evidence-based smoking treatment available to them and ways to initiate treatment (i.e., warm hand-off from a clinical provider).
  Arms: Enhanced Chronic Care
Behavioral: Standard Care — Standard Care involves one call per year. During the Standard Care call, participants will be encouraged to quit smoking, reminded of the cessation treatment available to them, and provided with a number to call should they become interested in treatment.
  Arms: Standard Care

SUMMARY:
This project will generate knowledge about the effectiveness of Enhanced Chronic Care, an intervention designed to enhance treatment use and smoking abstinence in Veterans who are initially unwilling to quit. Enhanced Chronic Care provides ongoing motivational interventions and interpersonal support designed to promote readiness to quit smoking. Enhanced Chronic Care will be compared with Standard Care (brief advice to quit once per year) on criteria that are of great clinical and public health importance: use of cessation treatment and smoking abstinence. It is expected that Enhanced Chronic Care will increase treatment use and smoking abstinence relative to Standard Care.

DETAILED DESCRIPTION:
This project will generate knowledge about the effectiveness of Enhanced Chronic Care, an intervention designed to enhance treatment use and smoking abstinence in Veterans who are initially unwilling to quit. Enhanced Chronic Care provides ongoing motivational interventions and interpersonal support designed to promote readiness to quit smoking. Enhanced Chronic Care will be compared with Standard Care (brief advice to quit once per year) on criteria that are of great clinical and public health importance: smoking treatment reach (use of cessation treatment) and abstinence. It is expected that Enhanced Chronic Care will increase treatment use and smoking abstinence relative to Standard Care.

The investigators will evaluate these interventions using a 2-arm randomized controlled trial. Veterans who smoke daily, but who are not willing to enter smoking cessation treatment, will be eligible to participate, with no obligation to quit smoking. Participants (N=500) will be randomized to one of the following treatments: 1) Enhanced Chronic Care (n=250) or 2) Standard Care (n=250). These intervention conditions will last 2 years to permit analysis of their cumulative impact on abstinence and treatment use

ELIGIBILITY:
Inclusion Criteria:

* Not willing to set a quit date in the next 30 days
* Report smoking an average of 4 or more cigarettes daily for at least six months
* Read, write, and speak English
* Be medically eligible to use nicotine replacement therapy
* If female, use an approved method of birth control if they use nicotine replacement therapy
* Agree to participate in the study
* Be at least 18 years old
* Be a Veteran

Exclusion Criteria:

* Unable to give informed, voluntary consent to participate
* Current use of any pharmacotherapy for smoking cessation not provided by the researchers during tobacco treatment
* Use of non-cigarette tobacco products as a primary form of tobacco use
* Incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
7-Day Point-Prevalence Abstinence | 2 years
  Participants who self-report no smoking for the past 7 days at the assessment endpoint (2-year follow-up) will be considered to meet criteria for 7-Day Point-Prevalence Abstinence. Participants who report any smoking in the past 7 days (at the 2 year follow-up) will be considered to be relapsed (smoking).

SECONDARY OUTCOMES:
Initiating at least 1 cessation treatment call | 2 years
  Cessation treatment use will be defined as making at least one treatment contact (initiating at least 1 cessation treatment call with reach coded as a binary outcome: use vs. no use).

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Megan Cook, PhD, Principal Investigator — William S. Middleton Memorial Veterans Hospital, Madison, WI
Locations (1):
- William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT04061720/ICF_000.pdf